CLINICAL TRIAL: NCT04194125
Title: Clinical Study of Radiopeptide 177Lu-DOTATOC in Combination With Capecitabine and Temozolomide in Advanced, Non-resectable and Progressive Neuroendocrine Tumors With Somatostatin Receptor Overexpression
Brief Title: Personalized CAPTEM Radiopeptide Therapy of Advanced, Non-resectable Neuroendocrine Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Warmia and Mazury (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Medical University of Warsaw (Other); The Diagnostic and Therapeutic Center Gammed; Poland (Unknown); National Center for Research and Development, Poland (Other)
Responsible Party: Principal Investigator, Jaroslaw B. Cwikla, MD, PhD, Professor UWM, Head of Department of Nuclear Medicine, University of Warmia and Mazury
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLNETS_2018
Record Dates: First submitted 2019-12-07; First posted 2019-12-11 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Neuroendocrine Tumors
Keywords: PRRT - Peptide Receptor Radionuclide Therapy; CAPTEM - Capecitabine-temozolomide; GET-NET - Gastro-Entero-Pancreatic Neuroendocrine Tumours; PFS - progression free survival; OS - overall survival
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-DOTATOC combined with CAPTEM (Experimental): * The therapy will include 4 courses (14 days per one) with 8-week intervals;
  * 177Lu-DOTATOC in doses from 5,55GBq up to 7,4 GBq will be administered i.v. up to four times at 10th day;
  * Concomitant amino acids will be given with each administration;
  * Capecitabine will be administrated for 14 days (twice a day) followed by Temozolomide at 10-14th days in each therapy sessions.
  Interventions: Drug: 177Lu-DOTATOC

INTERVENTIONS:
Drug: 177Lu-DOTATOC — Four administrations of 5,55GBq up to 7,4 GBq 177Lu-DOTATOC will be administered at 8-week intervals.

SUMMARY:
This is a non-randomized, phase II, open label study. The purpose of this study is to estimate Progression Free Survival (PFS) after treatment with Peptide Receptor Radionuclide Therapy (PRRT) 177Lu-DOTATOC standard dose (up to 4x7,4GBq 177Lu DOTATOC) in combination with capecitabine (CAP) and temozolomide (TEM) - CAPTEM.

Patients with advanced, non-resectable and/or progressive gastro-entero-pancreatic neuroendocrine tumors, GEP-NET, (G1, G2), in selected cases with high proliferation index (Ki-67> 20%, usually below 55%), NETG3, with overexpression of somatostatin receptor (SSTR positive) will be enrolled in the study.

DETAILED DESCRIPTION:
This is a non-randomized, phase II, open label study.

The purpose of this study is to:

• estimate Progression Free Survival (PFS) after treatment with Peptide Receptor Radionuclide Therapy (PRRT) 177Lu-DOTATOC standard dose (up to 4x7,4GBq 177Lu DOTATOC) in combination with capecitabine (CAP) and temozolomide (TEM) - CAPTEM.

Patients with advanced, non-resectable and/or progressive gastro-entero-pancreatic neuroendocrine tumors, GEP-NET according to WHO 2017 classification, (histological grade G1, G2), in selected cases patients with high proliferation index (Ki-67> 20%, usually below 55%), NETG3 - pancreatic, midgut neuroendocrine tumors and carcinoma of unknown primary (CUP). All with overexpression of somatostatin receptor (SSTR positive) based on somatostin receptor scintigraphy (SRS), will be enrolled in this study.

* evaluate the safety and tolerability of combination therapy using 177Lu-DOTATOC and CAPTEM.
* evaluate the health related quality of life (QoL) as measured by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-G.I.NET21 questionnaire.
* evaluate internal dosimetry, in a subset up to 20 patients, but at least 10 patients.
* explore the correlation of clinical efficacy outcomes with Somatostatin Receptor Scintigraphy (SRS) using 99mTc HYNICTOC (Tektordyt®) tumour uptake score.
* explore the correlation of clinical efficacy outcomes with the levels of some specific and non-specific biomarkers and gene transcripts analysis.
* compare the Time to Tumour Progression (TTP).

The schedule of treatment will include 4 courses; capecitabine (CAP), which will be administrated for 14 days with 8-week breaks, combined at 10th day with 177Lu-DOTATOC (PRRT - Peptide Receptor Radionuclide Therapy) in doses from 5,55GBq up to 7,4 GBq administered i.v. up to four times in every patient during whole therapy.

In selected patients, in those with only liver involvement or dominant liver bulky disease third and fourth administration of PRRT will be used intra-arterial administration (i.a.) via hepatic artery. The administered dose will be from 2.85 GBq up to 3.7GBq, up to two times per whole therapy, followed in each case of i.v. or i.a. PRRT by Temozolomide (TEM) p.o. administration, which will be given during 10-14th days in each therapy sessions.

Doses of PRRT could be modified due to clinical stage and laboratory parameters. Treatment will be discontinued in the case of a cumulative dose 29,6 GBq, corresponding to the radiation dose on the bone marrow below 2 Gy and cumulative dose on kidney below 23 Gy. In case of radiation dose on kidney above 23 Gy treatment will be interrupted.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old, male or female;
* All patients with histologically proven, well/moderate-differentiated G1/2 GEP-NET (according to WHO 2017 classification), with Ki-67 ≤20%, in selected cases patients with NETG3 will be included if there will be reported well/moderate morphological appearance but Ki-67>20% but less then Ki<30% (pancreatic, midgut NET and cancer with unknown primary (CUP)); and there will be high expression of somatostatin receptor seen in functional imaging utilized functional imaging 99mTc HYNICTOC or 68Ga DOTATATE or 68Ga DOTATOC;
* The presence of high expression of somatostatin receptors demonstrated on Somatostatin Receptor Imaging using 99mTc HYNICTOC (SPECT) or 68Ga DOTATATE or 68Ga DOTATOC (PET) scans, et least as uptake in not involved liver, Krenning >2;
* Non-resectable, advanced determined by an appropriately specialized surgeon or deemed not suitable for liver directed therapies where liver is the only site of disease;
* Performance status (PS) based on ECOG 0-2;
* Unresectable, advanced/metastatic progressive disease evaluated as clinical, biochemical, bad control symptoms of tumour hypersecretion or disease progression seen in imaging structural or functional;
* Parameteres of laboratory test:

  1. Morphology: Hb>10g/dl, PLT>75x103/ml, WBC> 2x103 /ml with ACN> 1.5x103/ml
  2. Adequate renal function (GFR>30 ml/min)*, creatinine <1.5 mg/dl
  3. Adequate liver function (Bilirubin <1.8 mg/dl, ALAT and ASPAT, AP <5 ULN (ULN - upper limit of normal) * The patient may be qualificated to supportive treatment if the patient's condition is stable.
* Life expectancy of at least 6 months;
* The tumor parameters that can be measured objectively as the size to be assessed in radiological studies on the basis of the RECIST 1.0 and RECIST 1.1;
* In the absence of the ability to measure tumor size based on RECIST criteria, they have tumor parameters that can be measured objectively as tumor markers determined in the blood or urine CgA, 5HIAA;
* Study treatment both planned and able to start within 28 days of inclusion;
* Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments;
* Signed, written informed consent.

Exclusion Criteria:

* Patients <18 years old;
* Coexistence of another cancer during recent 5 years, except cancers treated with curative intention and confirmed cured in follow-up with no or low risk of relapse;
* Allergy on somatostatin receptor analogues or capecitabine and temozolomide;
* Previous cytotoxic chemotherapy e.g. CAPTEM, and/or radiopeptide therapy PRRT;
* Pre-existing locoregional treatment such as radiomebolization (SIRspheres) or HDR brachytherapy under CT control, performed in the last 6 months;
* Uncontrolled metastases to the central nervous system, in the case of surgical and/or radiotherapeutic treatment, patients should remain on a stable dose of steroids for at least 2 weeks before enrollment, without deterioration of the general state associated with the presence of metastatic disease in the CNS;
* Poorly controlled concurrent medical illness. E.g. unstable diabetes with glycosylated hemoglobin (HbA1c> 9.0), the optimal glycaemic control should be achieved before starting trial therapy);
* Major surgery/surgical therapy for any cause within three months before starting trial therapy;
* Symptomatic heart failure NYHA class III or IV, congestive cardiac failure, myocardial infarction in the last 6 months, serious uncontrolled cardiac arrhythmia, unstable angina, or other serious cardiac problems;
* Patients with malabsorption or other gastrointestinal disorders that may interfere with the oral absorption of capecitabine and temozolomide (e.g. colitis ulcerosa, persistent nausea, vomiting, persistent diarrhea) not suitable for conservative treatment and no reaction to SST receptor analogs (Sandostatin LAR or Somatulina Autogel), malabsorption syndrome, short bowel syndrome after resection
* Active uncontrolled infection, including Hepatitis and Hepatitis, HIV, in the case of HCV and HBV infection, the patient can be included in the study confirming the suppression of viral replication and the patient remains on the correct therapeutic dose of antiviral drugs;
* Pregnant patients (a negative pregnancy test is required);
* Women of childbearing age must present a negative pregnancy test at the beginning of the study and must use double barrier to contraception. Women of childbearing age are defined as menopausal if they remain not menstrual for at least 1 year, or surgical sterilization or removal of the uterus before the start of the study;
* Breast-feeding female patients;
* Patients in a mental state who can't understand the nature, extent and possible consequences of participating in the study associated with radioisotope treatment, or there is evidence of a lack of cooperation by the patient;
* Exclusive clinical and laboratory findings that may compromise the patient's safety or reduce the chances of obtaining satisfactory data to achieve the goal (s) of the study;
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse;
* The patient may be included in the maintenance treatment if the patient's clinical condition is stable.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
PFS - Progression Free Survival | 3 years
  the time from the start of treatment date to the date of first observation of documented local recurrence, metastases or disease progression. Patients without progression at the time of analysis will be censored. The median PFS will be estimated.
  Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  CT or MRI tumour assessment will be used to response evaluation. CT/MRI tumour assessment will be performed before start of PRRT and then after 6+2 weeks after last PRRT session followed by 6 months intervals during first 3 years of follow-up, after that annually. The measurement of PFS will be calculated in months.

SECONDARY OUTCOMES:
OS - Overall Survival (time months) | 5 years
  Overall survival is defined as the time from the date of the start therapy to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off. The measurement of OS will be calculated in months.
Performance Status (PS) - evaluation criteria | 5 years
  Clinical response based on physical performance status (PS) using standard evaluation based on WHO/ECOG criteria. It will be assessed before each treatment cycle and then followed by 6 weeks after completion of therapy and then at three-month intervals. The measurement will be in the scale as follows: 0-asymptomatic, 1=symptomatic but completely ambulatory, 2=Symptomatic <50% in bed during the day, 3= Symptomatic >50% in bed during the day; 4=Bedbound; 5=Death.
Cancer Related Symptoms - assessment of clinical criteria | 5 years
  Clinical response based on potential relief in the initial phase before PRRT during and after PRRT. Items will be assessed, including: appetite, malaise, pain associated with the disease, nausea, vomiting, fever, wheezing and abdominal pain or any other symptoms of advanced cancer. All of the above will be assessed as yes / no. Intensity will be recorded in the quality assessment. It will be evaluated before treatment, before each treatment cycle, and then 6 weeks after the end of therapy, and then at three-month intervals. The measurement will be made in the qualitative data set and categorized as improvement, stabilization or disease progression.
Hormonal overproduction symptoms - assessment of clinical criteria | 5 years
  Hormonal response based on relief of symptoms of hormonal overproduction, which will be compare to clinical symptoms before PRRT, during and after PRRT during clinical follow-up. The presence of specific symptoms with hormone overproduction including: 1. Carcinoid syndrome (CS) - initial intensity of diarrhea and potential relief after PRRT (number per day), initial intensity of flushing and potential relief after PRRT (number per day). 2. Presence of heartburn in case of NET with ZES (Zollinger-Elisson syndrome) initial intensity and potential relief during PRRT and after finished PRRT during clinical follow-up. 3. Presence of hypoglycemia in case of NET with insulin overproduction (insulinoma), initial intensity of hypoglycemia before PRRT and potential relief after PRRT during clinical follow-up. The measurement will be made in a set of the qualitative data as improvement, stabilization or disease progression.
ORR - Objective Response Rate - evaluation criteria | 5 years
  The evaluation of objective response will be utilized by multiphase structural imaging before and after i.v. contrast enhancement (CT or MRI). The radiological response will be based on RECIST 1.0 using standard terminology of objective response, performed before start of PRRT and then after 6+2 weeks after last PRRT therapy followed by 6 months intervals during first 3 years of follow-up, after that annually. The measurement will be made in a set of quantitative data as partial response (PR), stable disease (SD) or disease progression (DP).
Safety Assessments - Laboratory Parameters - evaluation criteria: CTCAEs ver. 5.0 | 5 years
  Changes from Baseline in Hematology (WBC, RBC, platelets, haemoglobin), Blood chemistry (BUN, serum creatinine and creatinine clearance, uric acid, albumin, total bilirubin, AP, aspartate aminotransferase [AST/ASAT], alanine aminotransferase [ALT/ALAT], gamma-glutamyl transferase [γ-GT], [Na], [K], lactic dehydrogenase [LDH], glycosylated hemoglobin/hemoglobin A1c [glycoHb] and specific biomarkers Chromogranin-A (CgA) in the serum and 5-Hydroxyindoleacetic acid (5-HIAA) in the urine. The measurement will be made in a set of quantitative data, based on CTCAEs ver. 5.0 tep.cancer.gov/protocolDevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_5x7.pdf
Vital Signs - heart rate - physiological parameter | 5 years
  heart rate (beats per minute)
Systolic and diastolic blood pressure - physiological parameter | 5 years
  mmHg
BMI - Body Mass Index - physiological parameter | 5 years
  weight (kg), height (m) Body Mass Index (BMI kg/m2). The measurement will be made in a set of quantitative data
ECG - physiological parameter | 5 years
  ECG analysis during each therapy session and clinical follow-up, including: P Wave, QRS Complex, QT Interval. The measurement will be made in a set of quantitative data

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum Diagnostyczno-Lecznicze Gammed, Warsaw, Poland

REFERENCES:
- [Background] Strosberg JR, Fine RL, Choi J, Nasir A, Coppola D, Chen DT, Helm J, Kvols L. First-line chemotherapy with capecitabine and temozolomide in patients with metastatic pancreatic endocrine carcinomas. Cancer. 2011 Jan 15;117(2):268-75. doi: 10.1002/cncr.25425. Epub 2010 Sep 7. PMID 20824724
- [Background] Welin S, Sorbye H, Sebjornsen S, Knappskog S, Busch C, Oberg K. Clinical effect of temozolomide-based chemotherapy in poorly differentiated endocrine carcinoma after progression on first-line chemotherapy. Cancer. 2011 Oct 15;117(20):4617-22. doi: 10.1002/cncr.26124. Epub 2011 Mar 31. PMID 21456005
- [Background] Fine RL, Gulati AP, Krantz BA, Moss RA, Schreibman S, Tsushima DA, Mowatt KB, Dinnen RD, Mao Y, Stevens PD, Schrope B, Allendorf J, Lee JA, Sherman WH, Chabot JA. Capecitabine and temozolomide (CAPTEM) for metastatic, well-differentiated neuroendocrine cancers: The Pancreas Center at Columbia University experience. Cancer Chemother Pharmacol. 2013 Mar;71(3):663-70. doi: 10.1007/s00280-012-2055-z. Epub 2013 Jan 31. PMID 23370660
- [Background] Saif MW, Kaley K, Brennan M, Garcon MC, Rodriguez G, Rodriguez T. A retrospective study of capecitabine/temozolomide (CAPTEM) regimen in the treatment of metastatic pancreatic neuroendocrine tumors (pNETs) after failing previous therapy. JOP. 2013 Sep 10;14(5):498-501. doi: 10.6092/1590-8577/1589. PMID 24018594
- [Background] Peixoto RD, Noonan KL, Pavlovich P, Kennecke HF, Lim HJ. Outcomes of patients treated with capecitabine and temozolamide for advanced pancreatic neuroendocrine tumors (PNETs) and non-PNETs. J Gastrointest Oncol. 2014 Aug;5(4):247-52. doi: 10.3978/j.issn.2078-6891.2014.019. PMID 25083296
- [Background] Koumarianou A, Kaltsas G, Kulke MH, Oberg K, Strosberg JR, Spada F, Galdy S, Barberis M, Fumagalli C, Berruti A, Fazio N. Temozolomide in Advanced Neuroendocrine Neoplasms: Pharmacological and Clinical Aspects. Neuroendocrinology. 2015;101(4):274-88. doi: 10.1159/000430816. Epub 2015 Apr 29. PMID 25924937
- [Background] De Divitiis C, von Arx C, Grimaldi AM, Cicala D, Tatangelo F, Arcella A, Romano GM, Simeone E, Iaffaioli RV, Ascierto PA, Tafuto S; European Neuroendocrine Tumor Society (ENETS) Center of Excellence-Multidisciplinary Group for Neuroendocrine Tumors in Naples (Italy). Metronomic temozolomide as second line treatment for metastatic poorly differentiated pancreatic neuroendocrine carcinoma. J Transl Med. 2016 May 3;14(1):113. doi: 10.1186/s12967-016-0857-1. PMID 27142424
- [Background] Ramirez RA, Beyer DT, Chauhan A, Boudreaux JP, Wang YZ, Woltering EA. The Role of Capecitabine/Temozolomide in Metastatic Neuroendocrine Tumors. Oncologist. 2016 Jun;21(6):671-5. doi: 10.1634/theoncologist.2015-0470. Epub 2016 May 25. PMID 27226359
- [Background] Kwekkeboom DJ, de Herder WW, Kam BL, van Eijck CH, van Essen M, Kooij PP, Feelders RA, van Aken MO, Krenning EP. Treatment with the radiolabeled somatostatin analog [177 Lu-DOTA 0,Tyr3]octreotate: toxicity, efficacy, and survival. J Clin Oncol. 2008 May 1;26(13):2124-30. doi: 10.1200/JCO.2007.15.2553. PMID 18445841
- [Background] Cwikla JB, Sankowski A, Seklecka N, Buscombe JR, Nasierowska-Guttmejer A, Jeziorski KG, Mikolajczak R, Pawlak D, Stepien K, Walecki J. Efficacy of radionuclide treatment DOTATATE Y-90 in patients with progressive metastatic gastroenteropancreatic neuroendocrine carcinomas (GEP-NETs): a phase II study. Ann Oncol. 2010 Apr;21(4):787-794. doi: 10.1093/annonc/mdp372. Epub 2009 Oct 15. PMID 19833821
- [Background] Bodei L, Cremonesi M, Grana CM, Fazio N, Iodice S, Baio SM, Bartolomei M, Lombardo D, Ferrari ME, Sansovini M, Chinol M, Paganelli G. Peptide receptor radionuclide therapy with (1)(7)(7)Lu-DOTATATE: the IEO phase I-II study. Eur J Nucl Med Mol Imaging. 2011 Dec;38(12):2125-35. doi: 10.1007/s00259-011-1902-1. Epub 2011 Sep 3. PMID 21892623
- [Background] Hicks RJ, Kwekkeboom DJ, Krenning E, Bodei L, Grozinsky-Glasberg S, Arnold R, Borbath I, Cwikla J, Toumpanakis C, Kaltsas G, Davies P, Horsch D, Tiensuu Janson E, Ramage J; Antibes Consensus Conference participants. ENETS Consensus Guidelines for the Standards of Care in Neuroendocrine Neoplasia: Peptide Receptor Radionuclide Therapy with Radiolabeled Somatostatin Analogues. Neuroendocrinology. 2017;105(3):295-309. doi: 10.1159/000475526. Epub 2017 Apr 13. No abstract available. PMID 28402980
- [Background] Claringbold PG, Turner JH. Pancreatic Neuroendocrine Tumor Control: Durable Objective Response to Combination 177Lu-Octreotate-Capecitabine-Temozolomide Radiopeptide Chemotherapy. Neuroendocrinology. 2016;103(5):432-9. doi: 10.1159/000434723. Epub 2015 Jun 10. PMID 26065489
- [Background] Claringbold PG, Brayshaw PA, Price RA, Turner JH. Phase II study of radiopeptide 177Lu-octreotate and capecitabine therapy of progressive disseminated neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2011 Feb;38(2):302-11. doi: 10.1007/s00259-010-1631-x. Epub 2010 Oct 30. PMID 21052661